CLINICAL TRIAL: NCT01852591
Title: Exploration of Immune Response to Pneumococcal Conjugate Vaccine (PCV13) Administered Before and Early After Autologous Peripheral Stem Cell Transplant (Auto-PSCT) in Patients With Multiple Myeloma
Brief Title: Exploration of Immune Response to Early PCV13 Vaccination in Conjunction With Autologous Transplant
Acronym: PCV13
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MCC-16727
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma
Keywords: autologous transplant; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 13-valent pneumococcal vaccine; Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PCV 13 (Experimental): Pneumococcal conjugate vaccine (PCV 13), 0.5ml, 3 to 30 days prior to transplant and then again at 7-10 and 21-24 days after transplant
  Interventions: Biological: PCV 13

INTERVENTIONS:
Biological: PCV 13
  Other Names: Prevnar; pneumococcal conjugate vaccine

SUMMARY:
There is no study hypothesis. The purpose of this study is to see if the Pneumococcal conjugate vaccine (PCV13), when administered before and early after an autologous peripheral stem cell transplant will induce an immune response.

DETAILED DESCRIPTION:
This is a pilot study to determine the safety of PCV13 administered to patients with myeloma before and at +7-10 days and +21-24 days after autologous hematopoietic stem cell transplant; and,to quantify the immune response induced by PCV13 vaccination in patients with myeloma when administered before and early after autologous PSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed multiple myeloma
* Eligible for treatment with high dose melphalan based regimen and autologous peripheral stem cell transplant

Exclusion Criteria:

* Pregnant or lactating woman, as evaluated by serum testing within 24 hours of administration of the first vaccine
* HIV infection confirmed by nucleic acid testing (NAT), as evaluated during pre transplant testing
* Common variable immunodeficiency or other inherited systemic immunodeficiency syndrome
* Active central nervous system (CNS) malignancy
* Prior malignancy within 5 years of enrollment excluding non-melanoma skin cancer or cervical carcinoma after curative resection, not requiring chemotherapy.
* History of severe allergy (e.g., anaphylaxis) to any component of pneumococcal conjugate vaccine 7 (PCV7), PCV13, or any diphtheria-toxoid containing vaccine.
* Inclusion on a separate trial in which patients may be randomized or otherwise started on maintenance chemotherapies within the first 3 months of autologous transplantation
* Patients with significant psychiatric illness likely to affect compliance, as determined by the treating physician
* Active or uncontrolled infection
* Diffusing lung capacity oxygenation (DLCO) <50 %
* Left ventricular ejection fraction (LVEF) <40%
* Bilirubin >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Locke, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H.Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: H.Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org
- See also: Bone Marrow Transplantation advance online publication 12 October 2015; doi: 10.1038/bmt.2015.239 — http://www.nature.com/bmt/journal/vaop/ncurrent/full/bmt2015239a.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center between March 2013 and July 2014.
Groups:
- Experimental: PCV 13: Pneumococcal conjugate vaccine (PCV 13), 0.5ml, 3 to 30 days prior to transplant and then again at 7-10 and 21-24 days after transplant.
Period: Overall Study
Arm/Group | Experimental: PCV 13
Started | 8
Completed | 5
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Not Evaluable at Time of Analysis | 1

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | Experimental: PCV 13
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 61.625 [52 to 68]
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immune Response
Description: Positive response per test category. Post-vaccination result higher than pre-vaccination values for each test category criteria. Additional details are reported under Secondary Outcome Measures.
Time Frame: 30 Days Post Vaccine
Population: All evaluable participants.
Measure: Number; unit: participants
Arm/Group | Experimental: PCV 13
Number analyzed (Participants) | 5
participants
  CD4+CTV-IFN-gamma+, | 5
  CD8+CTV-IFN-gamma+, | 5
  CD8+CD107a+ | 5

2. Secondary Outcome: CD4+CTV-IFN-gamma+, Best Response Against Vaccine (CRM 197)
Description: Best CD4+ response against CRM197 at day +30 after transplant, utilizing flow cytometry for interferon-γ (IFN-gamma). Peripheral blood mononuclear cells were stained with cell trace violet (CTV) then incubated with CRM197 or vehicle control. Cells were then harvested and stained for flow cytometry.
Time Frame: 30 Days Post Vaccine
Population: All evaluable participants.
Measure: Number; unit: percentage of CD4 cells
Arm/Group | Experimental: PCV 13
Number analyzed (Participants) | 5
percentage of CD4 cells
  Highest % of CD4 cells Pre-vaccine | 0.051
  Best Response % of CD4 cells Day +30 | 40.7

3. Secondary Outcome: CD8+CTV-IFN-gamma+, Best Response Against Vaccine (CRM 197)
Description: Best CD8+ response against CRM197 at day +30 after transplant, utilizing flow cytometry for interferon-γ (IFN-gamma). Peripheral blood mononuclear cells were stained with cell trace violet then incubated with CRM197 or vehicle control. Cells were then harvested and stained for flow cytometry. Highest percentage increase of CD8 cells from pre-vaccine to Day + 30.
Time Frame: 30 Days Post Vaccine
Population: All evaluable participants.
Measure: Number; unit: percentage of CD8 cells
Arm/Group | Experimental: PCV 13
Number analyzed (Participants) | 5
percentage of CD8 cells
  Highest % of CD8 cells Pre-vaccine | 0.00
  Best Response % of CD8 cells Day +30 | 2.69

4. Secondary Outcome: CD8+CD107a+, Best Response Against Vaccine (CRM 197)
Description: Best CD8+ response against CRM197 at day +30 for CD107a. Peripheral Blood Mononuclear Cells (PBMCs) were incubated with CRM197, or control. Cells were harvested and stained for flow cytometry.
Time Frame: 30 Days Post Vaccine
Population: All evaluable participants.
Measure: Number; unit: percentage of CD8 cells
Arm/Group | Experimental: PCV 13
Number analyzed (Participants) | 5
percentage of CD8 cells
  Highest % of CD8 cells Pre-vaccine | 1.19
  Best Response % of CD8 cells Day +30 | 8.94

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Description: All participants who received treatment.
Arm/Group | Experimental: PCV 13
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: PCV 13 (N=7)
Cardiac disorders - Other, Orthostasis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Abdminal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: PCV 13 (N=7)
Headache (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fever (General disorders) | 5 (5)
Injection site reaction (General disorders) | 4 (9)
Edema limbs (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Other, Heartburn (Gastrointestinal disorders) | 1 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Papulopustular rash (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Hallucinations (Psychiatric disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibriliation (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes